CLINICAL TRIAL: NCT04391894
Title: A Randomized, Double-masked, Multicenter Study to Evaluate the Safety and Efficacy of ECF843 vs Vehicle in Subjects With Dry Eye Disease
Brief Title: A Study to Assess the Safety and Efficacy of ECF843 vs Vehicle in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CECF843A2201
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
Keywords: Dry Eye; Sjogrens; dry eye syndrome (DES); Keratoconjunctivitis sicca (KCS); keratitis; Xerophthalmia; Sjögren's Syndrome; Sjogren's Syndrome
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis Sicca; Keratitis; Xerophthalmia; Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- ECF843 0.45 mg/mL TID or vehicle (Part 1) (Experimental): ECF843 0.45 mg/mL TID or vehicle (Part 1)
  Interventions: Drug: ECF843; Other: ECF843 vehicle
- ECF843 0.15 mg/mL TID or vehicle (Part 1) (Experimental): ECF843 0.15 mg/mL TID or vehicle (Part 1)
  Interventions: Drug: ECF843; Other: ECF843 vehicle
- ECF843 vehicle TID (Part 1) (Placebo Comparator): ECF843 vehicle TID (Part 1)
  Interventions: Other: ECF843 vehicle
- ECF843 0.15 mg/mL BID or vehicle (Part 1) (Experimental): ECF843 0.15 mg/mL BID or vehicle (Part 1)
  Interventions: Drug: ECF843; Other: ECF843 vehicle
- ECF843 vehicle BID (Part 1) (Placebo Comparator): ECF843 vehicle BID (Part 1)
  Interventions: Other: ECF843 vehicle

INTERVENTIONS:
Drug: ECF843 — Topical ocular eye drop
  Arms: ECF843 0.15 mg/mL BID or vehicle (Part 1); ECF843 0.15 mg/mL TID or vehicle (Part 1); ECF843 0.45 mg/mL TID or vehicle (Part 1)
Other: ECF843 vehicle — Topical ocular eye drop

SUMMARY:
The study was planned to be conducted in 2 parts: Part 1 to determine the efficacy and safety of ECF843 vs vehicle, followed by Part 2 with additional exploratory assessments of ECF843 vs Vehicle. Both parts of the study included a double-masked study design, with randomization stratified for subjects with Sjogren's Syndrome.

DETAILED DESCRIPTION:
Part 1 of the study was a double-masked, randomized, parallel design in which participants were assigned to one of the following five treatment arms/groups in a ratio of 1:1:1:1:1.

* ECF843 0.45 mg/mL three times daily (TID) or vehicle
* ECF843 0.15 mg/mL TID or vehicle
* ECF843 vehicle TID
* ECF843 0.15 mg/mL twice daily (BID) or vehicle
* ECF843 vehicle BID The planned duration of double-masked treatment during Part 1 was 56 days. For subjects randomized to ECF843, the maximum drug exposure was up to 28 days. At some point during Part 1, all participants received vehicle.

The study was terminated after completion of Part 1 and Part 2 of the study was not therefore initiated.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment
* Adult male or female subjects 18 years of age or older
* At least 6 months history of dry eye disease in both eyes
* Must use, or feel the need to use, artificial tears/gels/lubricants on a regular basis
* Composite corneal fluorescein staining score >= 4 (modified National Eye Institute (NEI) scale) in at least one eye
* Schirmer score >= 1 and =< 10 mm after 5 minutes in at least one eye
* Patients with Sjögren's Syndrome must have dry eye

Exclusion Criteria:

* Ocular infection in either eye within 30 days prior to Screening
* Use of artificial tears, gels, lubricants within 4 hours of the Screening Visit
* Use of contact lenses in either eye within 14 days of Screening
* Uncontrolled ocular rosacea
* Clinically significant conjunctivochalasis in either eye
* Other Corneal conditions affecting the corneal structure
* Severe ocular conditions such as herpes, graft versus host disease, Stephen's Johnson Syndrome, sarcoidosis
* Currently active, or history of ocular allergies during the time of year the patient will be participating in the study
* Patients with current punctal plugs or punctal cauterization or occlusion
* Chronic medications (both over the counter and prescription) that have not been stable for at least 30 days prior to Screening.
* Use of Restasis®, Cequa®, or Xiidra® within 30 days prior to Screening
* Use of ocular, nasal, inhaled, or systemic corticosteroids within 30 days of Screening
* History of malignancy of any organ system within the past five years
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 718 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (52):
- United States (52):
  - Arizona Eye Center, Chandler, Arizona
  - Carrot Eye Center, Mesa, Arizona
  - Phoenix Eye Care and Dry Eye Ctr, Phoenix, Arizona
  - Milton Hom OD, Azusa, California
  - Orange County Opthamology Med Grp, Garden Grove, California
  - Dr Kent Small, Glendale, California
  - Global Research Management, Glendale, California
  - United Medical Research Institute, Inglewood, California
  - Harvard Eye Associates, Laguna Hills, California
  - North Valley Eye Medical Group, Mission Hills, California
  - The Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates Inc, Petaluma, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Sierra Clin Trials Rsch Org, Santa Ana, California
  - Vision Institute, Colorado Springs, Colorado
  - Advanced Research LLC, Deerfield Beach, Florida
  - Pinnacle Research Institute, Fort Lauderdale, Florida
  - Eye Associates Of Fort Myers, Fort Myers, Florida
  - Lee Shettle Eye & Hearing, Largo, Florida
  - Mid Florida Eye Center Pa, Mt. Dora, Florida
  - Kannarr Eye Care, Pittsburg, Kansas
  - The Eye Care Institute, Louisville, Kentucky
  - Tufts Medical Center, Boston, Massachusetts
  - Silverstein Eye Centers, Kansas City, Missouri
  - Moyes Eye Center, Kansas City, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Comprehensive Eye Care Limited, Washington, Missouri
  - NV Eye Surgery, Henderson, Nevada
  - AdvanceMed Clinical Research, Las Vegas, Nevada
  - Northern New Jersey Eye Institut PA, South Orange, New Jersey
  - Cornerstone Eye Care, High Point, North Carolina
  - Eye Care Assoc of Greater Cincinnati Inc, Cincinnati, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - Apex Eye Clinical Reserach, Mason, Ohio
  - Scott Christie Eye Care Associates, Cranberry Township, Pennsylvania
  - Bucci Laser Vision Institute, Wilkes-Barre Township, Pennsylvania
  - Vance Thompson Vision Hospital, Sioux Falls, South Dakota
  - Chattanooga Eye Institute, Chattanooga, Tennessee
  - University Eye Specialists, Maryville, Tennessee
  - Total Eye Care PA, Memphis, Tennessee
  - Toyos Clinic, Nashville, Tennessee
  - Advancing Vision Research LLC, Smyrna, Tennessee
  - Texan Eye P A, Austin, Texas
  - Intouch Clinical Research Center, Houston, Texas
  - Neuro Eye Clinical Trials Inc, Houston, Texas
  - Revolution Research, Lakeway, Texas
  - Parkhurst NuVision, San Antonio, Texas
  - Stacy R Smith MD PC, Salt Lake City, Utah
  - Southern Utah Medical Research, St. George, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Virginia Eye Consultants, Norfolk, Virginia
  - Periman Eye Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 53 sites in the USA.
Pre-assignment Details: Approximately 800 subjects were planned to be screened in Part 1 to have approximately 680 subjects randomized into the 56-day treatment period. A total of 970 subjects were screened, of which 558 subjects received randomized treatment.
Groups:
- ECF843 0.45 mg/mL TID (Part 1): ECF843 0.45 mg/mL ter in die/three times a day (TID) (Part 1)
- ECF843 0.15 mg/mL TID (Part 1): ECF843 0.15 mg/mL ter in die/three times a day (TID) (Part 1)
- ECF843 Vehicle TID (Part 1): ECF843 vehicle ter in die/three times a day (TID) (Part 1)
- ECF843 0.15 mg/mL BID (Part 1): ECF843 0.15 mg/mL bis in diem/twice a day (BID) (Part 1)
- ECF843 Vehicle BID (Part 1): ECF843 vehicle bis in diem/twice a day (BID) (Part 1)
Period: Overall Study
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1)
Started (All randomized treated subjects were included in Full Analysis Set 1 (FAS1) and Safety Set 1 (SAF1)) | 111 | 112 | 112 | 109 | 114
Completed | 107 | 111 | 108 | 107 | 111
Not Completed | 4 | 1 | 4 | 2 | 3
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 0 | 1
Not completed — Unsatisfactory Therapeutic effect | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1) | Total
Number analyzed (Participants) | 111 | 112 | 112 | 109 | 114 | 558
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.7 (13.68) | 60.6 (13.64) | 62.1 (12.89) | 62.9 (13.51) | 62.7 (13.04) | 62.0 (13.33)
Age, Customized [Number; unit: Participants]
  < 65 years | 56 | 60 | 55 | 49 | 59 | 279
  >= 65 years | 55 | 52 | 57 | 60 | 55 | 279
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 89 | 86 | 82 | 83 | 423
  Male | 28 | 23 | 26 | 27 | 31 | 135
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 20 | 17 | 12 | 19 | 83
  Not Hispanic or Latino | 96 | 92 | 95 | 97 | 95 | 475
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 3 | 4 | 2 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 16 | 17 | 24 | 15 | 12 | 84
  White | 89 | 88 | 85 | 90 | 99 | 451
  More than one race | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Sjogren's Syndrome status [Count of Participants; unit: Participants] — Status of Sjogren's syndrome was based on history of diagnosis.
  Participants
    Yes | 4 | 4 | 4 | 2 | 5 | 19
    No | 107 | 108 | 108 | 107 | 109 | 539

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Symptom Assessment in Dry Eye (SANDE) Score
Description: The SANDE uses a 100 mm visual analog scale (VAS) and asks the subject to score frequency and severity of their ocular discomfort over the past 24 hours by putting a vertical mark on two separate horizontal scoring lines. The frequency scoring line utilizes the anchors of 'Rarely' to 'All the Time', while the severity scoring line utilizes the anchors of 'Very Mildly' to 'Very Severely uncomfortable'. The SANDE questionnaire was completed through an electronic diary by the subject at the Screening Visit(s) of Part 1, and thereafter every evening before bedtime during the study. The overall SANDE score was calculated by taking the square root of the product of the frequency of symptoms score and the severity of symptoms score. The SANDE scale ranged from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount of dry eye symptoms. Negative change from baseline indicates improvement.
Time Frame: Up to 28 days (Baseline (BL) to end of randomized treatment)
Population: Full Analysis Set 1 including subjects with a value at both Baseline and post-baseline visit. Baseline is defined as the last available value collected prior to or on the first administration of randomized study treatment.
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1)
Number analyzed (Participants) | 111 | 112 | 112 | 109 | 114
Score on scale | -6.0 (1.86) | -8.1 (1.85) | -4.9 (1.85) | -1.8 (1.91) | -6.1 (1.84)
Statistical Analysis 1: Comparison: ECF843 0.45 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; p = 0.585, Mixed Models Analysis; Least Squares Mean (LS Mean) = -1.1, 95% CI 2-sided [-5.0 to 2.8], Standard Error of Mean 2.01
Statistical Analysis 2: Comparison: ECF843 0.15 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; p = 0.107, Mixed Models Analysis; Least Squares Mean (LS Mean) = -3.2, 95% CI 2-sided [-7.01 to 0.7], Standard Error of Mean 2.00
Statistical Analysis 3: Comparison: ECF843 0.15 mg/mL BID (Part 1) vs ECF843 Vehicle BID (Part 1); Test type: Superiority; p = 0.033, Mixed Models Analysis; Least Squares Mean (LS Mean) = 4.3, 95% CI 2-sided [0.3 to 8.3], Standard Error of Mean 2.02

2. Primary Outcome: Part 1: Change From Baseline in Composite Corneal Fluorescein Staining Score
Description: The degree of staining was based on the Corneal Fluorescein Modified NEI Scale. Each of the five regions (central (C), superior (S), inferior (I), temporal (T), and nasal (N)) were graded based on a scale of 0 to 4, with higher scores suggestive of higher degrees of corneal staining. After entry of the scores per region, the total or composite (sum) score for each eye was automatically calculated (maximum score = 20/eye). A (+1) was added to the sum score for any eye with the presence of filaments.
Time Frame: Up to 28 days (Baseline (BL) to end of randomized treatment)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score on scale
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1)
Number analyzed (Participants) | 111 | 112 | 112 | 109 | 114
Score on scale | -1.1 (0.30) | -1.0 (0.30) | -0.9 (0.30) | -1.0 (0.31) | -1.1 (0.30)
Statistical Analysis 1: Comparison: ECF843 0.45 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; p = 0.605, Mixed Models Analysis; Least Squares Mean (LS Mean) = -0.2, 95% CI 2-sided [-0.8 to 0.4], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: ECF843 0.15 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; p = 0.646, Mixed Models Analysis; Least Squares Mean (LS Mean) = -0.1, 95% CI 2-sided [-0.7 to 0.5], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: ECF843 0.15 mg/mL BID (Part 1) vs ECF843 Vehicle BID (Part 1); Test type: Superiority; p = 0.847, Mixed Models Analysis; Least Squares Mean (LS Mean) = 0.1, 95% CI 2-sided [-0.5 to 0.7], Standard Error of Mean 0.31

3. Secondary Outcome: Part 1: Change From Baseline in Central Corneal Fluorescein Staining
Description: The degree of staining was based on the Corneal Fluorescein Modified NEI Scale. Central region was graded based on a scale of 0 to 4, with higher scores suggestive of higher degrees of corneal staining.
Time Frame: Up to 28 days (Baseline (BL) to end of randomized treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1)
Number analyzed (Participants) | 107 | 111 | 110 | 108 | 110
Score on scale | -0.2 (0.80) | -0.3 (0.78) | -0.2 (0.83) | -0.2 (0.65) | -0.2 (0.74)
Statistical Analysis 1: Comparison: ECF843 0.45 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: ECF843 0.15 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.11
Statistical Analysis 3: Comparison: ECF843 0.15 mg/mL BID (Part 1) vs ECF843 Vehicle BID (Part 1); Test type: Superiority; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.09

4. Secondary Outcome: Part 1: Change From Baseline in Inferior Corneal Fluorescein Staining
Description: The degree of staining was based on the Corneal Fluorescein Modified NEI Scale. Inferior region was graded based on a scale of 0 to 4, with higher scores suggestive of higher degrees of corneal staining.
Time Frame: Up to 28 days (Baseline (BL) to end of randomized treatment)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1)
Number analyzed (Participants) | 107 | 111 | 110 | 108 | 110
Score on scale | -0.2 (0.75) | -0.3 (0.85) | -0.2 (0.89) | -0.2 (0.98) | -0.6 (1.06)
Statistical Analysis 1: Comparison: ECF843 0.45 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; Mean Difference (Net) = -0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: ECF843 0.15 mg/mL TID (Part 1) vs ECF843 Vehicle TID (Part 1); Test type: Superiority; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.12
Statistical Analysis 3: Comparison: ECF843 0.15 mg/mL BID (Part 1) vs ECF843 Vehicle BID (Part 1); Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [0.1 to 0.6], Standard Error of Mean 0.14

5. Secondary Outcome: Part 1: Percentage of Participants With Ocular and Non-ocular Treatment Emergent Adverse Events (AEs)
Description: The number of treatment emergent ocular and non-ocular adverse events was reported categorically: Mild, Moderate, Severe.
  Treatment emergent adverse events (TEAEs) are adverse events started after the first administration of randomized study treatment or events present prior to start of the randomized treatment but increased in severity based on preferred term.
Time Frame: Up to 28 days (Baseline (BL) to end of randomized treatment)
Population: Safety Set 1
Measure: Count of Participants; unit: Participants
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1)
Number analyzed (Participants) | 111 | 112 | 112 | 109 | 114
Participants
  Ocular treatment emergent adverse events: number analyzed (Participants) | 5 | 10 | 5 | 2 | 7
  Ocular treatment emergent adverse events: Mild | 5 | 10 | 4 | 2 | 7
  Ocular treatment emergent adverse events: Moderate | 0 | 0 | 1 | 0 | 0
  Ocular treatment emergent adverse events: Severe | 0 | 0 | 0 | 0 | 0
  Non-ocular treatment emergent adverse events: number analyzed (Participants) | 5 | 6 | 1 | 3 | 4
  Non-ocular treatment emergent adverse events: Mild | 4 | 5 | 0 | 1 | 3
  Non-ocular treatment emergent adverse events: Moderate | 1 | 1 | 1 | 2 | 1
  Non-ocular treatment emergent adverse events: Severe | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 28 days (Baseline (BL) to end of randomized treatment)
Description: All safety evaluations were carried out on the Safety Set 1 (SAF1). The SAF1 included all participants who received at least one dose of study treatment in Part 1. The analysis was done according to the study treatment received, where treatment received was defined as the actual randomized treatment if the subject took at least one dose of that treatment or the first treatment received if the randomized treatment was never received.
Arm/Group | ECF843 0.45 mg/mL TID (Part 1) | ECF843 0.15 mg/mL TID (Part 1) | ECF843 Vehicle TID (Part 1) | ECF843 0.15 mg/mL BID (Part 1) | ECF843 Vehicle BID (Part 1)
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/112 | 0/112 | 0/109 | 0/114
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/112 | 1/112 | 0/109 | 1/114
Other Adverse Events (participants affected / at risk) | 9/111 | 15/112 | 5/112 | 5/109 | 12/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ECF843 0.45 mg/mL TID (Part 1) (N=111) | ECF843 0.15 mg/mL TID (Part 1) (N=112) | ECF843 Vehicle TID (Part 1) (N=112) | ECF843 0.15 mg/mL BID (Part 1) (N=109) | ECF843 Vehicle BID (Part 1) (N=114)
Pelvic mass (General disorders) | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ECF843 0.45 mg/mL TID (Part 1) (N=111) | ECF843 0.15 mg/mL TID (Part 1) (N=112) | ECF843 Vehicle TID (Part 1) (N=112) | ECF843 0.15 mg/mL BID (Part 1) (N=109) | ECF843 Vehicle BID (Part 1) (N=114)
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 1 | 1 | 0 | 0 | 0
Chalazion (Eye disorders) | 0 | 0 | 1 | 0 | 2
Conjunctival deposit (Eye disorders) | 0 | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 2
Corneal erosion (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 1 | 2 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 2 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 0 | 0 | 1 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0 | 0 | 0
Glare (Eye disorders) | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Instillation site pain (General disorders) | 1 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 3 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/94/NCT04391894/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT04391894/SAP_001.pdf